CLINICAL TRIAL: NCT04407455
Title: Inter-rater Reliability in Determining Chewing Performance Level in Children
Brief Title: Determining Chewing Performance Level in Children
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SELEN SEREL ARSLAN, Principal Investigator, Hacettepe University
Other Study IDs: Chewing performance level
Record Dates: First submitted 2020-05-25; First posted 2020-05-29 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Chewing Problem

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with cerebral palsy: Children who will be referred to pediatric dentistry above the age of 2 years.
  Interventions: Diagnostic Test: Karaduman Chewing Performance Scale
- Children with typical development: Children who will be referred to pediatric dentistry above the age of 2 years.
  Interventions: Diagnostic Test: Karaduman Chewing Performance Scale

INTERVENTIONS:
Diagnostic Test: Karaduman Chewing Performance Scale — For chewing evaluation, children will be asked to bite and chew a standardized biscuit. Each chewing evaluation will be scored according to the KCPS.

SUMMARY:
The study will investigate to verify whether pediatric dentists could determine chewing performance level by using Karaduman Chewing Performance Scale in children.

DETAILED DESCRIPTION:
The KCPS was developed by physical therapists who had expertise in pediatric swallowing disorders. This scale could be used as a practical tool to define chewing disorders as a common language for professionals due to its quick and easy to use features. However, its reliability in other professions has not been verified. The study will investigate to verify whether pediatric dentists could determine chewing performance level by using Karaduman Chewing Performance Scale in children.

ELIGIBILITY:
Inclusion Criteria:

* Typical developing children
* Children with cerebral palsy (CP)
* Above the age of 2 years

Exclusion Criteria:

* Children who were under the age of 2 years
* Who used any medicine and/or oral appliances that may affect chewing performance
* Who had a previous evaluation of chewing function and received any chewing training

Ages: 2 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: Typical developing children and children with cerebral palsy (CP) who will be referred to pediatric dentistry above the age of 2 years.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Karaduman Chewing Performance Scale | 2 months
  The Karaduman Chewing Performance Scale is a 5 level ordinal scale between 0 to 4. Level 0 indicates Normal chewing, level 4 means No biting and chewing. Higher levels mean worse chewing performance level.

CONTACTS AND LOCATIONS:
Overall Officials: SELEN SEREL ARSLAN, Principal Investigator — Hacettepe University
Locations (1):
- Hacetttepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Serel Arslan S, Ozsin Ozler C, Demir N, Ozturk S, Uzamis Tekcicek M, Karaduman AA. Pediatric dentists can determine chewing performance level in children. Clin Oral Investig. 2021 Aug;25(8):5043-5048. doi: 10.1007/s00784-021-03815-w. Epub 2021 Feb 2. PMID 33528675